CLINICAL TRIAL: NCT07093242
Title: Functional Epigenetic Optimization Through Biofrequency-Guided Nutrition: A Randomized Controlled Trial
Brief Title: Epigenetic Optimization Through Biofrequency Nutrition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Cell wellbeing (Unknown)
Responsible Party: Principal Investigator, David Manzano, David Manzano Sánchez, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UALBIO2025/010
Record Dates: First submitted 2025-07-09; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Nutrition Habits; Biomarkers / Hair; Epigenetic
Keywords: Biofrequency analysis; young athletes; nutritional intervention; nutritional biomarkers; mediterranean diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Nutritional Follow-Up (Experimental): Participants in this group receive a genetic hair analysis and a personalized nutritional follow-up based on the results. The aim is to assess whether the nutritional intervention modifies relevant genetic or biochemical markers after the intervention period.
  Interventions: Behavioral: Personalized Nutritional Follow-Up
- Control Group - Results Only (No Intervention): Participants in this group receive a genetic hair analysis and are provided with the results only, without any nutritional follow-up. This group serves as a comparison to evaluate the effect of the nutritional intervention in the experimental group.

INTERVENTIONS:
Behavioral: Personalized Nutritional Follow-Up — Participants in the experimental arm will receive a individual nutritional follow-up based on their epigenetic hair analysis results. This includes dietary guidance, recommendations tailored to genetic markers, and periodic consultations with a nutritionist over 4 weeks and continuous availability to clarify doubts via email . The aim is to evaluate changes in genetic expression or health biomarkers after the intervention period.
  Arms: Experimental Group - Nutritional Follow-Up

SUMMARY:
Biomarker-based nutrition has demonstrated superior efficacy compared to population-level approaches in improving health outcomes. Biofrequency analysis, a non-invasive technique based on the detection of electromagnetic vibrational patterns in hair follicles, offers a promising avenue for rapid functional assessment of nutritional status and epigenetic signals without reliance on blood or urine sampling. First, to evaluate the effect of a 90-day biofrequency-guided nutritional intervention on functional epigenetic status, as reflected in changes in the optimization report generated by the S-Drive system; second, to assess changes in adherence to the Mediterranean diet, anthropometric indicators, movement behaviors, and psychological well-being. Methods: In this randomized controlled trial, adults from a Sport Team from Region of Murcia (Spain) will be allocated to an experimental group receiving individualized lifestyle recommendations based on S-Drive biofrequency analysis and to a control group with no intervention. Participants in the experimental arm will apply tailored dietary guidance over 90 days. Conclusion: This study will generate foundational evidence on the utility of biofrequency technology for precision nutrition. If positive, the findings may inform scalable, low-risk strategies for personalized dietary interventions in preventive and community health settings.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Active member of a registered athletics club.
* Willingness to provide a hair sample for genetic analysis.
* Ability to understand and sign the informed consent form.
* Commitment to complete the nutritional follow-up (for the intervention group) and to respond to pre- and post-intervention questionnaires.

Exclusion Criteria:

* Prior medical diagnosis of a genetic disorder affecting nutritional metabolism.
* Current use of nutritional supplements or special diets prescribed for medical reasons.
* Participation in another clinical or nutritional study during the intervention period.
* Pregnancy or breastfeeding at the time of enrollment.
* Inability to attend baseline or post-intervention assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in biofrequency-derived epigenetic markers related to nutritional metabolism | baseline and after 12-weeks post-intervention
  This outcome evaluates the correlation between the nutritional intervention and functional epigenetic status, assessed through the S-Drive optimization report. The measurement tool is the S-Drive system (Cell Wellbeing, Germany), a non-invasive device that analyzes resonance frequency patterns from hair follicle samples using proprietary bioinformatic algorithms. The report classifies physiological function into 12 domains related to nutritional metabolism (e.g., micronutrients, oxidative stress, circulatory function), assigning ordinal values to each: "not flagged" (0), "to be considered" (1), "advisable" (2), or "priority" (3). Two derived quantitative variables will be analyzed: (1) the number of domains classified as "priority" (unit: count, range: 0-12), and (2) the cumulative optimization score summing the ordinal ratings (unit: score, range: 0-36). These biofrequency will be used to assess within-subject changes and between group correlations from baseline to 90-day follow-up.
Adherence to the Mediterranean Diet measured by the 14-item PREDIMED questionnaire | Baseline and after 12 weeks of intervention
  This outcome assesses adherence to the Mediterranean dietary pattern using the validated 14-item PREDIMED questionnaire (PREvención con DIeta MEDiterránea). Each item is scored as 0 (non-compliance) or 1 (compliance), for a total score ranging from 0 to 14. Higher scores indicate better adherence. The unit of measurement is the total PREDIMED score. A score ≥9 is considered high adherence. This variable will be measured at baseline and after the 90-day intervention to evaluate correlations between the individualized nutritional guidance and improvement in diet quality in the experimental group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: David Manzano Sánchez, Principal Investigator — Universidad de Almeria

IPD SHARING:
Plan to Share IPD: Undecided
The participants' data will be anonymized to protect confidentiality and will not be shared with other researchers

REFERENCES:
- See also: Related Info — https://www.cell-wellbeing.es

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT07093242/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT07093242/ICF_001.pdf